CLINICAL TRIAL: NCT07073599
Title: The Effect of Breast and Gynecological Cancer Education Using Creative Drama Method on Midwifery Students' Awareness: A Randomized Controlled Trial
Brief Title: Increasing Midwifery Students' Awareness of Breast and Gynecological Cancers Using Creative Drama Method
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zülbiye demir barbak, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Creative drama in midwifery
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Creative Drama
Keywords: Creative drama; Breast and gynecological cancers; Midwifery students; Awareness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive routine training and no action will be taken.
- Experimental Group (Experimental): Students in the intervention group will be given a creative drama session. This will evaluate the impact of creative drama training on breast and gynecological cancer awareness.
  Interventions: Other: Creative Drama Education

INTERVENTIONS:
Other: Creative Drama Education — This study is a pre-test/post-test controlled experimental design aimed at evaluating the effectiveness of creative drama education on awareness of breast and gynecological cancers.
  Students in the intervention group will receive creative drama-based training structured and implemented by the researcher. This training is designed to increase awareness of breast and gynecological cancers.
  The effectiveness of the training will be assessed by comparing participants' awareness levels before and after the intervention. For this purpose, the following data collection tools will be used:
  Personal Information Form Breast Cancer Awareness Scale Gynecological Cancers Awareness Scale The impact of the creative drama education on the awareness levels of students in the intervention group regarding breast and gynecological cancers will be evaluated through statistical analysis.
  Arms: Experimental Group

SUMMARY:
The aim of this study is to raise awareness among midwifery students, who are a part of the female population and a professional group that plays a critical role in the early diagnosis of these types of cancer, which are of critical importance for women's health, through an active education method such as drama.

DETAILED DESCRIPTION:
The study will involve 50 volunteer midwifery students between the ages of 18 and 35 studying at the Faculty of Health Sciences. Students will be randomized and assigned to experimental and control groups. Awareness levels of breast and gynecological cancers in both groups will be determined. Students in the intervention group will be administered a creative drama exercise. Data will be collected using a Personal Information Form, the Breast Cancer Awareness Scale, and the Gynecological Cancer Awareness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35,
* Not having any health problems,
* Agreeing to participate in the study,

Exclusion Criteria:

* Students who are under 18 or over 35 years old.
* Students who do not voluntarily agree to participate in the study will not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Personel Information Form | Baseline
  The researcher will prepare a form based on literature information and will question the students' sociodemographic characteristics.
Gynecological Cancers Awareness Scale | Baseline and up to 4 weeks
  To assess women's knowledge levels about gynecological cancers, Dal and Ertem developed the Gynecological Cancer Awareness Scale (GCAAS) in 2017. The scale consists of 41 questions and four subscales. 10. The scale can only be applied to women. The Cronbach's alpha value of the scale is 0.944. Questions 20-41 of the scale determine "Awareness of Routine Check-up and Perception of Serious Illness in Gynecological Cancers," and the Cronbach's alpha value of this subscale is 0.979. Questions three through 11 of the scale determine "Awareness of Gynecological Cancer Risks," and the Cronbach's alpha value of this subscale is 0.843. Questions 14-19 of the scale determine "Awareness of Prevention of Gynecological Cancers," and the Cronbach's alpha value is 0.778. The first and second questions of the scale, as well as the 12th and 13th questions, determine "Early Diagnosis and Information Awareness in Gynecological Cancers," and the Cronbach's Alpha value is 0.708.
Breast Cancer Awareness Scale | Baseline and up to 4 weeks
  The scale was developed by Rakkapao et al. (2016) for the early detection and prevention of breast cancer. It is easy to use and was designed as a self-report tool that allows researchers and practitioners to better understand women's breast cancer awareness levels. The original scale consists of five factors and 35 items. Adapted to our language by Altuntuğ et al. in 2021, the scale obtained a five-factor structure with 29 items. The subdimensions of the scale were found to have good internal consistency. The Cronbach's alpha internal consistency coefficients for the subdimensions of the scale were 0.87 for Knowledge of Risk Factors, 0.88 for Knowledge of Signs and Symptoms, 0.81 for Breast Cancer Prevention Attitudes, 0.78 for Barriers to Breast Screening, and 0.61 for Health Behavior Related to Breast Cancer Awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Zülbiye DEMİR BARBAK, 1, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Health Sciences, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erci B, Karabulut N. Appraising the self-assessed support needs of Turkish women with breast cancer. Eur J Cancer Care (Engl). 2007 Mar;16(2):137-43. doi: 10.1111/j.1365-2354.2006.00721.x. PMID 17371422
- See also: Validity and Reliability — https://pubmed.ncbi.nlm.nih.gov/17371422/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17371422/